CLINICAL TRIAL: NCT05828693
Title: Efficacy of Systemic Stress Prevention Via Application SysLife© for Companies: A Randomized Controlled Feasibility Study
Brief Title: Systemic Stress Prevention Via Application SysLife© for Companies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Sysba solutions GmbH (Unknown); Murtfeldt Kunststoffe GmbH & Co. KG (Unknown)
Responsible Party: Principal Investigator, Christina Hunger-Schoppe, Chair for clinical psychology and psychotherapy, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SysLife©
Record Dates: First submitted 2022-12-12; First posted 2023-04-25 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stress, Psychological; Stress, Systemic; Application
Keywords: Stress management; Application, App; Prevention; Systemic therapy
MeSH Terms: conditions — Stress, Psychological; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Use of the SysLife© application, with 2-, 4-, 6- and 8-month follow-up.
  Interventions: Behavioral: SysLife©
- Waiting group with subsequent intervention (Other): Use of the SysLife© application after 4-month waiting period, with 2- and 4-month follow-up.
  Interventions: Behavioral: SysLife©, as intervention after closing the RCT-design

INTERVENTIONS:
Behavioral: SysLife© — Use of the SysLife© application, with 2-, 4-, 6- and 8-month follow-up.
  Arms: Experimental group
Behavioral: SysLife©, as intervention after closing the RCT-design — Use of the SysLife© application after 4-month waiting period, with 2- and 4-month follow-up.
  Arms: Waiting group with subsequent intervention

SUMMARY:
The purpose of this study is to investigate the efficacy of systemic stress prevention via SysLife© application in a prospective, interventive, balanced, monocentric, explanatory pilot randomized controlled trial (RCT), with participants' subjective stress experience as the primary endpoint.

Research Question: Which implementations are necessary, based on the experience from this pilot RCT, to ensure the quality of a subsequent confirmatory RCT?

Hypothesis: We expect improvement of participants' subjective stress experience, goal achievement, systemic functioning in private and organisational social systems while using the SysLife© application.

DETAILED DESCRIPTION:
Background: Systemic prevention serves the prophylaxis of disease and/or illness, and/or damage to health. For social subsystems such as professional teams, there however still is a lack of effective preventive or health-promoting interventions. With the Prevention Act introduced in 2015 (Social Security Code, Germany: § 20 para. 1 SGB V), prevention now has to address the social context of people's everyday life as well ("setting/life-world approach"). Positive changes in terms of reduced stress perception or acute exposition to stress factors are supposed to be accompanied by improved systemic, psychological and physical well-being. This RCT will investigate the efficacy of the systemic stress prevention program SysLife© application.

Methods: This prospective, interventive, balanced, monocentric, explanatory pilot RCT compares an experimental group (n = 19) receiving SysLife© application with a control group (n = 19) with subsequent intervention, i.e. the SysLife@ application 4 months after the experimental group. The primary endpoint is the participants' subjective stress experience.

The data collection encompasses 5 measurement points: t1, i.e. baseline for the experimental group; t2: 2-month follow-up; t3: 4-month follow-up for the experimental group and baseline for the control group; t4: 6-month follow-up for the experimental group and 2-month follow-up for the control group; t5: 8-month follow-up for the experimental group and 2-month follow-up for the control group).

This allows for the calculation of trends considering the potential efficacy of the SysLife© application in the RCT design on the one hand (n = 19, 2-study arm approach), and in a cumulative study (n = 38, 1-study arm approach).

Research Question: Which implementations are necessary, based on the experience from this pilot RCT, to ensure the quality of a subsequent confirmatory RCT?

Hypothesis: We expect improvement of participants' subjective stress experience, goal achievement, systemic functioning in private and organisational social systems while using the SysLife© application.

Questionnaires: Stress and Coping Inventory (SCI); Trier Stress Inventory (TICS); Experience in Social Systems (EXIS), Goal Attainment Scaling (GAS). Further items: demographic data, use of additional health care interventions, user behavior and effect of the SysLife© application.

Discussion: To the best of our knowledge, this will be the first prospective, interventive, balanced, monocentric, explanatory pilot RCT comparing SysLife© application with a waiting group. For study purposes, it is a challenge to implement SysLife© application in organizational contexts such as teams: systemic prevention is an innovative health-promoting approach which is not (yet) covered by the German health insurance companies; the SysLife© application is an innovative program in digital health management with high flexibility how to approach it while being standardized in its structure; though companies are increasingly interested in health-promoting interventions for their employees, they are sparing considering the investment of time and financial resources in occupational health care.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 18 years
* Interest in active use of the SysLife© application
* Knowledge of German at native language level or the ability to use German language independently (at least B-level)
* Only persons capable of giving consent will be included in the study
* Written consent to participate after information about the study

Exclusion Criteria:

* No written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline stress and coping at 4 months | baseline, 4-month follow-up
  Stress and Coping Inventory (SCI; Satow, 2012): Self-report measure to assess psychological and physical stress symptoms; Likert scale: 1 = not modified (positive), 7 = very strongly modified (negative)
Change from baseline chronic stress at 4 months | baseline, 4-month follow-up
  Trier Inventory on Chronic Stress (TICS; Schulz, Schlotz & Becker, 2004): Self-report measure to assess chronic stress; Likert scale: 0 = never (positive), 4 = very often (negative)

SECONDARY OUTCOMES:
Goal Attainment Scaling (GAS; Grosse Holtforth & Grawe, 2002) | baseline, 2-month follow-up, 4-month follow-up, 6-month follow-up, 8-month follow-up
  Self-report measure to assess participants' previously set goals and their achievement; Visual analogue scale: 0% = not reached at all, 100% = fully achieved
Experience in Social Systems (EXIS; Hunger et al., 2017) | baseline, 2-month follow-up, 4-month follow-up, 6-month follow-up, 8-month follow-up
  Self-report measure to assess systemic functioning in private and organizational social systems; Likert scale: 1 = not at all (negative), 6 = fully (positive)
Stress and Coping Inventory (SCI; Satow, 2012) | baseline, 2-month follow-up, 4-month follow-up, 6-month follow-up, 8-month follow-up
  Self-report measure to assess psychological and physical stress symptoms; Likert scale: 1 = not modified (positive), 7 = very strongly modified (negative)
Trier Inventory on Chronic Stress (TICS; Schulz, Schlotz & Becker, 2004) | baseline, 2-month follow-up, 4-month follow-up, 6-month follow-up, 8-month follow-up
  Self-report measure to assess chronic stress; Likert scale: 0 = never (positive), 4 = very often (negative)
Frequency of application use | baseline, 2-month follow-up, 4-month follow-up, 6-month follow-up, 8-month follow-up
  Program registration of user frequency; 0-1/week = infrequent use; 2-3/week = moderate use; 4-5/week = frequent use; 6-7/week = very frequent use

CONTACTS AND LOCATIONS:
Overall Officials: Christina Hunger-Schoppe, Prof. Dr., Study Director — University of Witten/Herdecke
Locations (1):
- Witten/Herdecke University, Witten, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunger C, Bornhauser A, Link L, Geigges J, Voss A, Weinhold J, Schweitzer J. The Experience in Personal Social Systems Questionnaire (EXIS.pers): Development and Psychometric Properties. Fam Process. 2017 Mar;56(1):154-170. doi: 10.1111/famp.12205. Epub 2016 Feb 8. PMID 26858173
- [Background] Barth, I., Immel, N. & Hunger-Schoppe, C. (2023). Systemische Prävention. [in print, Publisher: Kohlhammer]
- [Background] Satow, L. (2012). Stress and Coping Inventory (SCI). available under: http://www.drsatow.de/tests/stress-und-coping-inventar/
- [Background] Schulz, P., Schlotz, W. & Becker, P. (2004). Trier Inventory for Chronic Stress. Göttingen: Hogrefe.
- [Background] Grosse M, Grawe K. BERN INVENTORY OF TREATMENT GOALS: PART 1. Development and First Application of a Taxonomy of Treatment Goal Themes. Psychother Res. 2002 Mar 1;12(1):79-99. doi: 10.1080/713869618. PMID 22471333